CLINICAL TRIAL: NCT01819389
Title: Low-dose Nilotinib and Imatinib Combination in Chronic Myeloid Leukemia Patients, With Failure, Suboptimal Response or Treatment Intolerance.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, David Gomez Almaguer, MD, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE12-019
Record Dates: First submitted 2012-10-26; First posted 2013-03-27 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Leukemia, Myeloid, Chronic, BCR-ABL Positive
Keywords: Chronic myeloid leukemia; suboptimal response; imatinib; nilotinib
MeSH Terms: conditions — Leukemia; Bronchiolitis Obliterans Syndrome; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate; nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Imatinib and nilotinib combination (Experimental): All patients will receive treatment as follows: imatinib 100 mg tablets, 200 mg daily for 6 months; and nilotinib 150 mg capsule, 300 mg daily for 6 months.
  Interventions: Drug: Imatinib and Nilotinib

INTERVENTIONS:
Drug: Imatinib and Nilotinib
  Other Names: Gleevec; Tasigna

SUMMARY:
The purpose of this study is to determine if low-dose imatinib and nilotinib combination, will improve treatment results in CML patients with failure, suboptimal response or intolerance to imatinib therapy.

The hypothesis is that with low-dose imatinib and nilotinib combination, major molecular response will be achieved in patients not previously obtained with imatinib monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* CML patients with failure or suboptimal response to imatinib therapy according to criteria established by the European Leukemia Net (ELN)
* Patients with grade II or higher adverse events.
* CML patients not suitable for stem cell transplantation.

Exclusion Criteria:

* Patients in blast crisis.
* Pregnant women
* Patients without a contraception method.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-10; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Major molecular response | 6 months
  Major molecular response will be evaluated with quantitative Real time polymerase chain reaction assay (RT-PCR)for BCR/ABL at 6 months.

SECONDARY OUTCOMES:
Drugs adverese effects | 6 months
  Patients will be evaluated every four weeks to identify possible adverse effects of drugs administered.

OTHER OUTCOMES:
Adherence | 6 months
  Every month adherence will be assessed with a questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Servicio de Hematologia, Hospital Universitario "José E. Gonzalez", Monterrey, Nuevo León, Mexico

REFERENCES:
- [Background] Schoffski P, Reichardt P, Blay JY, Dumez H, Morgan JA, Ray-Coquard I, Hollaender N, Jappe A, Demetri GD. A phase I-II study of everolimus (RAD001) in combination with imatinib in patients with imatinib-resistant gastrointestinal stromal tumors. Ann Oncol. 2010 Oct;21(10):1990-1998. doi: 10.1093/annonc/mdq076. Epub 2010 May 27. PMID 20507881
- [Background] Gomez-Almaguer D, Tarin-Arzaga L, Cantu-Rodriguez O, Ceballos-Lopez A. More about imatinib and nilotinib combination therapy in chronic myeloid leukemia. Acta Haematol. 2013;129(1):18-9. doi: 10.1159/000342455. Epub 2012 Sep 12. No abstract available. PMID 22986736
- [Background] Zhu GR, Ji O, Ji JM, Zhang YC, Wu Y, Yu H, Jiang PJ, Shen Q. Combining nilotinib and imatinib improves the outcome of imatinib-resistant blast phase CML. Acta Haematol. 2012;127(3):152-5. doi: 10.1159/000333107. Epub 2012 Jan 27. PMID 22286512
- [Derived] Gomez-Almaguer D, Saldana-Vazquez R, Tarin-Arzaga L, Herrera-Rojas MA, Vazquez-Mellado de Larracoechea A, Cantu-Rodriguez OG, Gutierrez-Aguirre CH, Jaime-Perez JC. Combination of low-dose imatinib plus nilotinib for the treatment of chronic-phase chronic myeloid leukaemia after imatinib failure. Hematology. 2016 Aug;21(7):411-4. doi: 10.1080/10245332.2015.1119369. Epub 2016 Feb 16. PMID 26871197